CLINICAL TRIAL: NCT06363370
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Safety and Efficacy of Human Interferon α1b Inhaled Solution in the Treatment of Respiratory Syncytial Virus Lower Respiratory Tract Infection in Children.
Brief Title: Human Interferon α1b Inhalation Solution Against Respiratory Syncytial Virus in Children With Lower Respiratory Tract Infections
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kexing Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KXZY-GB05-201
Record Dates: First submitted 2024-04-07; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Human interferon α1b Inhalation Solution （4ug/kg） (Experimental): Participants will receive Human interferon α1b Inhalation Solution 4ug/kg twice daily for no more than 7 days.
  Interventions: Drug: Human interferon α1b Inhalation Solution
- Human interferon α1b Inhalation Solution（6ug/kg） (Experimental): Participants will receive Human interferon α1b Inhalation Solution 6ug/kg twice daily for no more than 7 days.
  Interventions: Drug: Human interferon α1b Inhalation Solution
- Inhalation Solution Placebo (Placebo Comparator): Participants will receive Placebo twice daily for no more than 7 days.
  Interventions: Drug: Inhalation Solution Placebo

INTERVENTIONS:
Drug: Human interferon α1b Inhalation Solution — Participants will receive Human interferon α1b Inhalation Solution
  Arms: Human interferon α1b Inhalation Solution （4ug/kg）; Human interferon α1b Inhalation Solution（6ug/kg）
Drug: Inhalation Solution Placebo — Participants will receive Inhalation Solution Placebo
  Arms: Inhalation Solution Placebo

SUMMARY:
To evaluate the efficacy and safety of interferon α1b (GB05) in the treatment of children under 2 years of age with respiratory syncytial virus infection.

DETAILED DESCRIPTION:
The study has been divided into two parts, 60 subjects will be randomly assigned to the 4μg/kg dose group or 6μg/kg dose group or the blank control group, to receive nebulized GB05 therapy, twice daily for no more than 7 days. After comprehensive evaluation of effectiveness and safety, and confirmation of the optimal dose, the sample size will be re-calculated to enter the second part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. 2 months ≤ age ≤ 2 years of age (including the correction age of premature babies, after the correction of the monthly age = (Current Date-birth date)-[(37 weeks-fetal age)/4], gender is not limited;
2. Comply with the following diagnostic criteria:

1) RSV real -time reversal transcript polymerase chain reaction (RT PCR) positive, or quantitative QPCR detection; Show the positive of RSV infection; 2) Cough and/or asthma, lung auspicious pitch and/or wet sounds; 3) Chest imaging examination shows the dot -shaped shadow and/or thick lung texture/slightly/more and/or emphysema and/or the signs of inflammation around the bronchial.

3. Signing the informed consent of the child's disease distance within 72 hours (cough, breathing, fever); 4. The severity of the condition of capillary bronchitis is moderate or severe; 5. The parents of the child, or the legal guardian, or the legal guardians have fully understood the relevant information of this experiment and the possible benefits and risks of the subject's expectations, and agreed that the child to participate in this experiment and voluntarily signed the informed consent.

Exclusion Criteria:

1. There is a history of drug allergies (interferon products, related solutions formula components, etc.), or those with a history of specific allergies (asthma, based on the "eczema area and severity index" (EASI for short) scoring method as severe eczema, etc.), Or those who are diagnosed by doctors clearly diagnose (such as allergies to two or more drugs, food and pollen);
2. Do not tolerate atomization inhalation to the administrator or suffer from severe oral and/or maxillofacial deformities, which affects the use of atomization inhalation;
3. Those who have genetic metabolic diseases;
4. A child with other respiratory pathogen infections (judgment based on the test results of respiratory pathogen)；
5. Any disabled drugs (disabled drugs include interferon, Libavarin and the drug instructions within 72 hours before the medication are expected to specify the Chinese medicines with antiviral effects, etc.) and within 24 hours before the administration of administration Children with sugar hormones used in inhalation and body;
6. There are severe cardiovascular (such as severe congenital heart disease, myocardial disease), the history of liver, kidney, and hemophilia.
7. There is a history of autoimmune diseases, such as autoimmune hemolytic anemia, thyroid autoimmune disease, ulcerative colitis, mixed connective tissue disease, dermatitis, etc.;
8. Those who are accompanied by basic diseases such as lung, bronchium, bronchial dysplasia;
9. Candid's with functional disorders and lesions with epilepsy or other central nervous system, such as meningitis, toxic or hypoxic encephalopathy;
10. During the filter, it is accompanied by severe diarrhea, moderate malnutrition, anemia, and blood system disease;
11. During the screening, the thoracic effusion, pydion and pus, and pus, etc.;
12. Merce able goose sores suspected mold infection during screening；
13. The laboratory inspection is abnormal during screening:1) White blood cell count>14x109/L (or normal value of normal value) or neutral granulocyte ratio> 70%, and researchers comprehensively judge suspects as merging bacterial infections;2) Excisibility of liver function test: Alanine aminotransferase (ALT) or permine aminamidase (AST)> The upper limit of the normal value is 2 times, or the total biliary erythrin> 1.5 times the upper limit of the normal value;3) Blood routine abnormalities: white blood cell count <3.5X109/L and/or platelet count≤100x109/L；
14. Extremely irritable, drowsiness, coma, or those who may need ventilator to assist breathing;
15. After the history of the history of the disease, the child known (or the mother who is younger than 6 months old) is HIV -positive, or the researcher is highly suspected of being HIV -positive;
16. In the random 30 days before the randomly participated in any drug clinical trial or those who used research drugs;
17. Volunteers may not be able to complete this study or researchers who believe that they are not suitable for participating in this clinical trial due to various reasons.

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 322 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Wang bronchiolitis score chanced by percentage from baseline | day 5
  The Wang bronchiolitis score consists of four sections (respiratory rate, stridor, respiratory muscle depression, general symptoms), and the severity of the patient's condition is from low to high on a scale of 0 to 12 on the scale. A score of < 5 indicates that the patient is mild, a score of 5-9 indicates that the patient is moderately ill, and a score of ≥9 indicates that the patient is severe.
Wang bronchiolitis score chanced by percentage from baseline | day 1 to day of last administration (except day 5)
  The Wang bronchiolitis score consists of four sections (respiratory rate, stridor, respiratory muscle depression, general symptoms), and the severity of the patient's condition is from low to high on a scale of 0 to 12 on the scale. A score of < 5 indicates that the patient is mild, a score of 5-9 indicates that the patient is moderately ill, and a score of ≥9 indicates that the patient is severe.
Wang bronchiolitis score of 0 in proportion | day 5
  The Wang bronchiolitis score consists of four sections (respiratory rate, stridor, respiratory muscle depression, general symptoms), and the severity of the patient's condition is from low to high on a scale of 0 to 12 on the scale. A score of < 5 indicates that the patient is mild, a score of 5-9 indicates that the patient is moderately ill, and a score of ≥9 indicates that the patient is severe.
Wang bronchiolitis score total score < 5 points | day 5
  The Wang bronchiolitis score consists of four sections (respiratory rate, stridor, respiratory muscle depression, general symptoms), and the severity of the patient's condition is from low to high on a scale of 0 to 12 on the scale. A score of < 5 indicates that the patient is mild, a score of 5-9 indicates that the patient is moderately ill, and a score of ≥9 indicates that the patient is severe.
Wang bronchiolitis score, the first time the total score reaches < 5 points | day 5
  The Wang bronchiolitis score consists of four sections (respiratory rate, stridor, respiratory muscle depression, general symptoms), and the severity of the patient's condition is from low to high on a scale of 0 to 12 on the scale. A score of < 5 indicates that the patient is mild, a score of 5-9 indicates that the patient is moderately ill, and a score of ≥9 indicates that the patient is severe.

SECONDARY OUTCOMES:
RSV viral load | From predose to 120 hours postdose
  qPCR test

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Capital Institute of Pediatrics, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No